CLINICAL TRIAL: NCT00689234
Title: Diaphragm Plication in Adults With Phrenic Nerve Paralysis: a Randomised Controlled Study
Brief Title: Diaphragm Plication in Adults With Phrenic Nerve Paralysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Marc Decramer, Prof. Dr., KU Leuven
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B32220083458 (no sponsor)
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Phrenic Nerve Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): At time of inclusion randomised in the "no intervention" arm (the subjects will be re-evaluated 6 months later and will get intervention at that time (cross-over protocol)
  Interventions: Procedure: diaphragm plication 6 months after inclusion
- B (Active Comparator): At time of inclusion the subject get the intervention
  Interventions: Procedure: diaphragm plication at time of inclusion

INTERVENTIONS:
Procedure: diaphragm plication 6 months after inclusion — thoracotomy
  Arms: A
Procedure: diaphragm plication at time of inclusion — thoracotomy
  Arms: B

SUMMARY:
The purpose of the study is to investigate the impact of unilateral or bilateral diaphragm plication in a prospective randomised controlled way on symptoms, pulmonary function including gas exchange, respiratory muscle strength, exercise capacity and breathing during sleep in patients with proven uni- or bilateral phrenic nerve paralysis present for at least 1 year without any evidence of spontaneous recovery.

ELIGIBILITY:
Inclusion Criteria:

* Uni- or bilateral diaphragmatic paralysis due to phrenic nerve paralysis present for at least 1 year
* With reduced VC, at least in supine position and no significant change in VC for at least 6 months
* At the time of randomisation symptomatic patient, defined by one of the following symptoms: not able to sleep in supine position or exertional dyspnoea

Exclusion Criteria:

* No informed consent obtained
* Other disease that may interfere with the evaluation of pulmonary function or the exercise capacity: COPD, parenchymal lung disease on the thoracic X-ray, documented ischemic heart disease or left heart failure, active rheumatological disease, severe orthopaedic problems,....
* Abnormal neuromuscular clinical investigation (apart from diaphragmatic dysfunction) and/or abnormal electromyography of the limbs compatible with generalized neuromuscular disease
* Known diseases resulting in abnormal blood coagulation
* Proven oncological origine of the phrenic nerve paralysis
* Age below 18 yrs old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Dyspnea | 6 months after inclusion
  Functional outcome measured by dyspnea score
Dyspnea | 12 months after inclusion
  Functional outcome measured by dyspnea score
Exercise capacity | 6 months after inclusion
  Functional outcome measured by exercise testing
Exercise capacity | 12 months after inclusion
  Functional outcome measured by exercise testing

SECONDARY OUTCOMES:
Pulmonary function | 6 months after inclusion
  Measurement of pulmonary function
Pulmonary function | 12 months after inclusion
  Measurement of pulmonary function
Sleep | 6 months after inclusion
  Polysomnography evaluation
Sleep | 12 months after inclusion
  Polysomnography evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Gasthuisberg Divisionof Pulmonology, Leuven, Belgium